CLINICAL TRIAL: NCT02105831
Title: Skeletal Muscle Perfusion With LVAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan R. Lindner, MD, Professor of Medicine, Oregon Health and Science University
Other Study IDs: CEU in LVAD
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Heart Failure
Keywords: left ventricular assist device; contrast ultrasound; perfusion imaging
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CEU skeletal muscle perfusion imaging: Heart failure with LVAD Contrast ultrasound skeletal muscle perfusion imaging
  Interventions: Other: Contrast ultrasound skeletal muscle perfusion imaging

INTERVENTIONS:
Other: Contrast ultrasound skeletal muscle perfusion imaging — 1. Contrast ultrasound perfusion imaging will be performed in patients in whom LVAD will be placed for clinical indications of severe heart failure.

SUMMARY:
Advanced heart failure (when the heart pump fails) is associated with symptoms such as shortness of breath and extreme fatigue. Some of these symptoms are simply due to failure of the pump, however abnormal regulation of blood flow to the muscles of the body is also a potential mechanism. Left ventricular assist devices are mechanical pumps used to compensate for patients with failing hearts either as a bridge to heart transplant or as long term therapy. Whether or not these pumps improve muscle flow and whether this is a determinant in the improvement of symptoms is unknown. Understanding how skeletal muscle and heart perfusion is altered in heart failure patients before and after implantation of an LVAD could provide further insight into the beneficial effects of this therapy.

Specific Aims:

1. To evaluate skeletal muscle and heart perfusion studies before and after LVAD implantation
2. To compare functional status with degree of skeletal muscle perfusion.

DETAILED DESCRIPTION:
Methods:

Thirty patients deemed to be candidates for LVAD from either outpatient heart failure clinic or inpatient cardiology service will be studies. Skeletal muscle perfusion imaging using standard of care ultrasound technology will be performed prior to LVAD implant and then 3 months post implant. Functional status by six minute walk test and specialized stress test will be assessed at 3 months post implant.

ELIGIBILITY:
Inclusion Criteria:

* patients deemed to be candidates for a LVAD

Exclusion Criteria:

* severe peripheral artery disease
* skeletal muscle disorder
* severe congenital heart disease
* pregnancy
* patients <18 yo

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Heart failure patients being referred for LVAD
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-02-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle perfusion on contrast enhanced ultrasound | 3 months
  Skeletal muscle perfusion will be quantified:
  1. Prior to LVAD placement
  2. 3 months post LVAD placement

SECONDARY OUTCOMES:
6 minute walk test | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States